CLINICAL TRIAL: NCT01944423
Title: Enhancing Panic and Smoking Reduction Treatment With D-Cycloserine
Acronym: DCS/PSRT
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Jasper A. Smits, Principal Investigator, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R34DA034658 (NIH)
Record Dates: First submitted 2013-09-10; First posted 2013-09-17 (Estimated); Results first posted 2021-05-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Nicotine Addiction; Panic Attack
MeSH Terms: conditions — Tobacco Use Disorder; Panic Disorder | interventions — Cycloserine; Sugars; Nicotine Replacement Therapy; Transdermal Patch; Nicotine; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PSRT_DCS (Experimental): Individuals in this condition will receive 7 weeks of panic and smoking reduction treatment (PSRT) and one pill of d-cycloserine (DCS) one hour prior to sessions 3, 4, and 5 (i.e., 3 single doses). Participants will also be given nicotine replacement therapy as part of PSRT (i.e., the patch).
  Interventions: Drug: d-cycloserine; Drug: Nicotine replacement therapy; Behavioral: Panic and Smoking Reduction Treatment
- PSRT_PBO (Placebo Comparator): Individuals in this condition will receive 7 weeks of panic and smoking reduction treatment (PSRT) and one pill placebo dose one hour prior to sessions 3, 4, and 5 (i.e., 3 single doses). Participants will also be given nicotine replacement therapy as part of PSRT (i.e., the patch).
  Interventions: Drug: Pill Placebo; Drug: Nicotine replacement therapy; Behavioral: Panic and Smoking Reduction Treatment

INTERVENTIONS:
Drug: d-cycloserine — d-cycloserine is a medication thought to be associated with fear extinction.
  Other Names: d-cycloserine; DCS
  Arms: PSRT_DCS
Drug: Pill Placebo
  Other Names: sugar pill
  Arms: PSRT_PBO
Drug: Nicotine replacement therapy — All participants will receive Nicoderm CQ®, 24-hour transdermal nicotine patches and will be educated about the use of the patch at the session immediately prior to quit date. They will be instructed to apply one patch daily, beginning on quit date (week 5). Participants will use the 3-step tapering Nicoderm process (21-mg, 14-mg, and 7-mg). This regimen has been used in previous trials with a similar formulation of the patch (Fiore, 2000). A meta-analysis found no differences in outcome between 16- or 24-hour patches (Fiore et al., 1994). Participants who continue to smoke or lapse after quit day will not be instructed to discontinue the patch until their smoking level reaches 4 cigarettes/day for 4 days. Smokers who lapse during treatment will be encouraged to set a new quit date and continue their cessation attempt.
  Other Names: patch, NRT, nicoderm,
Behavioral: Panic and Smoking Reduction Treatment — PSRT incorporates elements of standard smoking cessation treatment (i.e., counseling plus NRT) with procedures for reducing panic and enhancing tolerance to withdrawal sensations. Written therapist and patient manuals will be used and followed at all times to ensure standardized delivery of the treatment. Interventions that uniquely focus on addressing panic, fears and intolerance of anxiety, bodily-related sensations, and affect-relevant withdrawal symptoms include: (1) interoceptive exposure; (2) corrective information about anxiety and cognitive interventions designed to teach patients alternatives to catastrophic misinterpretations of the sensations and their feared consequences; and (3) situational exposure.
  Other Names: PSRT, CBT, cognitive behavioral therapy, panic reduction, smoking cessation

SUMMARY:
The purpose of the current study is to evaluate the efficacy of d-cycloserine in augmenting treatment of smoking cessation for individuals with panic attacks. The investigators hypothesize that individuals receiving DCS (versus those receiving placebo) will evidence greater smoking abstinence rates and decreased panic symptoms after receiving a combined CBT-based treatment for smokers with panic attacks.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ages 18-65 capable of providing informed consent
* Willing and able to provide informed consent, attend all study visits and comply with the protocol
* Daily smoker for at least one year
* Currently smoke an average of at least 8 cigarettes per day
* Report a motivation to quit smoking in the next month of at least 5 on a 10-point scale
* Evidence of panic attack within the past year and endorsement of smoking as an emotion regulation strategy (i.e., score at least a 78 on the SAEQ).

Exclusion Criteria:

* Subjects who do not use smoking as an emotion regulation strategy
* Current diagnosis of a psychotic, eating, developmental or bipolar disorder
* Significant suicide risk as determined by structured interview
* Pregnant women, lactating women, and women of childbearing potential who are not using medically accepted forms of contraception (e.g., IUD, oral contraceptives, barrier devices, condoms and foam, or implanted progesterone rods stabilized for at least 3 months).
* Psychoactive substance abuse or dependence (excluding nicotine dependence) within the past 6 months
* Current use of isoniazid or ethionamide compounds
* A history of significant medical condition and/or be deemed as currently unhealthy in the context of a complete physical examination
* Limited mental competency and the inability to give informed, voluntary, written consent to participate
* Current use of any pharmacotherapy or psychotherapy for smoking cessation not provided by the researchers during the quit attempt
* Concurrent psychotherapy initiated within three months of baseline, or ongoing psychotherapy of any duration directed specifically toward treatment of anxiety or mood disorder other than general supportive therapy initiated at least 3 months prior to the study
* Use of other tobacco products
* Plans to move outside of the immediate area in the next six months
* Insufficient command of the English language

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

REFERENCES:
- [Derived] Smits JAJ, Zvolensky MJ, Otto MW, Piper ME, Baird SO, Kauffman BY, Lee-Furman E, Alavi N, Dutcher CD, Papini S, Rosenfield B, Rosenfield D. Enhancing panic and smoking reduction treatment with D-Cycloserine: A pilot randomized clinical trial. Drug Alcohol Depend. 2020 Mar 1;208:107877. doi: 10.1016/j.drugalcdep.2020.107877. Epub 2020 Jan 22. PMID 32004998

RESULTS

PARTICIPANT FLOW:
Groups:
- PSRT_PBO: Individuals in this condition will receive 7 weeks of panic and smoking reduction treatment (PSRT) and one pill placebo dose one hour prior to sessions 3, 4, and 5 (i.e., 3 single doses). Participants will also be given nicotine replacement therapy as part of PSRT (i.e., the patch).
  Pill Placebo
Period: Overall Study
Arm/Group | PSRT_DCS | PSRT_PBO
Started | 27 | 26
End of Treatment | 21 | 20
1-month Follow-up | 22 | 19
4-month Follow-up | 19 | 16
Completed | 19 (6-month follow-up) | 17 (6-month follow-up)
Not Completed | 8 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PSRT_DCS | PSRT_PBO | Total
Number analyzed (Participants) | 27 | 26 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 26 | 53
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.19 (12.37) | 36.64 (12.85) | 35.91 (12.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 37
  Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 27 | 23 | 50
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 26 | 23 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 27 | 26 | 53

OUTCOME MEASURES:

1. Primary Outcome: Smoking Abstinence
Description: Smoking status will be assessed at baseline and each of the follow-up assessments using point prevalence abstinence (PPA) measures verified with carbon monoxide and saliva cotinine.
Time Frame: Assessed from week 3-29, week 29 reported
Population: Intent to treat analysis
Measure: Number; unit: percentage of participants
Arm/Group | PSRT_DCS | PSRT_PBO
Number analyzed (Participants) | 27 | 26
percentage of participants | 8.25 | 12.35
Statistical Analysis 1: Comparison: PSRT_DCS vs PSRT_PBO; Test type: Superiority; two-phase growth curve model — p=ns 2-sided; Logit difference (final values) = 0.64, 95% CI 2-sided [-2.25 to 0.97], Standard Error of Mean 0.82

2. Secondary Outcome: Anxiety Sensitivity Mechanistic Target
Description: Anxiety sensitivity was assessed using the Anxiety Sensitivity Index-3, which is an 18 item measure of fear of bodily sensations. Participants rated their concern regarding the possible negative consequences of internal anxiety-related sensations. Scores range from 0-72, with higher scores indicated greater sensitivity to bodily sensations (worse outcome).
Time Frame: Assessed from week 3-29, week 7 reported (end of treatment)
Population: Intent to treat analysis
Measure: Mean (Standard Deviation); unit: unstandardized units
Arm/Group | PSRT_DCS | PSRT_PBO
Number analyzed (Participants) | 27 | 26
unstandardized units | 15.37 (10.38) | 17.80 (13.77)
Statistical Analysis 1: Comparison: PSRT_DCS vs PSRT_PBO; At end-of-treatment; Test type: Superiority; p = .038, two-phase growth curve model — 2-sided; Mean Difference (Final Values) = 2.43, 95% CI 2-sided [0.25 to 7.94], Standard Error of Mean 1.87

3. Secondary Outcome: Panic Symptoms Mechanistic Target
Description: Panic disorder severity scale is a 7-item measure assessing the severity of seven features of panic: frequency of panic attacks, distress during panic attacks, anticipatory anxiety, agoraphobic fear and avoidance, interoceptive fear and avoidance, impairment of work functioning, and impairment of social functioning. Items are rated on a five-point Likert scale ranging from 0 (none) to 4 (extreme), with a total possible score of 28. Higher scores indicate greater severity and impairment.
Time Frame: Assessed from week 3-29, week 29 reported (6-month follow-up)
Population: Intent to treat analysis
Measure: Mean (Standard Deviation); unit: unstandardized units
Arm/Group | PSRT_DCS | PSRT_PBO
Number analyzed (Participants) | 27 | 26
unstandardized units | 5.36 (6.96) | 5.40 (5.93)
Statistical Analysis 1: Comparison: PSRT_DCS vs PSRT_PBO; At 6 month follow-up; Test type: Superiority; p = .003, two-phase growth curve model — 2-sided; Mean Difference (Final Values) = 3.21, 95% CI 2-sided [1.15 to 5.26], Standard Error of Mean 1

ADVERSE EVENTS:
Time Frame: Adverse event data was collected at each in-person appointmnet during the course of the study (baseline appointment through the 6-month follow-up).
Arm/Group | PSRT_DCS | PSRT_PBO
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/26
Other Adverse Events (participants affected / at risk) | 2/27 | 3/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PSRT_DCS (N=27) | PSRT_PBO (N=26)
Chipped back bone (General disorders) | 0 (0) | 1 (1) — Chipped bone in back reported at follow-up appointment. The event was deemed unrelated to study procedures.
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1) — Pericarditis reported at follow-up appointment. The event was deemed unrelated to study procedures.
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) — Participant reported elevated anxiety symptoms after 1st administration study medication. Deemed possibly related to study procedures and medication was discontinued.
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Participant was diagnosed with anemia during follow-up. AE was unlikely to be related to study procedures.
Migraine (General disorders) | 1 (1) | 0 (0) — Participant reported a migraine at follow-up appointment. AE was unlikely to be related to study procedures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-06-07): https://cdn.clinicaltrials.gov/large-docs/23/NCT01944423/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-07): https://cdn.clinicaltrials.gov/large-docs/23/NCT01944423/SAP_001.pdf